CLINICAL TRIAL: NCT07189832
Title: Bleomycin Intralesional Injections of Cystic Hygromas in Pediatric Patients
Brief Title: Bleomycin Intralesional Injections of Cystic Hygromas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Sarah Arafat, Lecturer, Delta University for Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 025081962
Record Dates: First submitted 2025-09-22; First posted 2025-09-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2024-09

CONDITIONS: Lymphatic Malformations
Keywords: Bleomycin, Cervico-facial, Cystic Hygroma, Lymphatic Malformation
MeSH Terms: conditions — Lymphatic Abnormalities; Lymphangioma, Cystic | interventions — Injections, Intralesional

STUDY DESIGN:
Intervention Model Description: pediatric patients of age up to 12 years having Cervicofacial cystic hygromas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intralesional Injections (Experimental): Bleomycin Intralesional Injections
  Interventions: Procedure: Intralesional Injections

INTERVENTIONS:
Procedure: Intralesional Injections — Intralesional Injections

SUMMARY:
Thirty pediatric patients with cystic hygromas participated in this study. The cystic fluid was aspirated from the cystic hygroma, and the lesion was simultaneously injected with Bleomycin. Then, the lesion was re-injected at 4-week intervals until satisfactory results were obtained. Clinical response was evaluated as complete response (> 90% reduction of lesion size), marked improvement (>70% reduction of lesion size), moderate improvement (40 - 70% reduction of lesion size), slight improvement (< 40%), and no response (< 10% reduction of lesion size).

DETAILED DESCRIPTION:
A total of 30 pediatric patients of age up to 12 years having Cervicofacial cystic hygromas (macrocystic lymphatic malformations) were chosen from the vascular anomalies clinic in Cairo University Specialized Pediatric Hospital (CUSPH). Diagnosis was accomplished by taking history from parents, clinical examination, and confirmed by ultrasonography (USG) and\or magnetic resonance imaging (MRI) for deep lesions.

The procedure was explained in simple, clear words to the parents of each infant/child before the study, and an informed written consent was signed by each parent, containing treatment benefits, potential risks as outlined in the principles of Helsinki Declaration. Each infant/child was treated and followed up for 12 months after the last BLM intralesional injection.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Cervicofacial cystic hygromas (macrocystic lymphatic malformations) Pediatric patients from age 1 month to 12 years, recruited from the vascular anomalies clinic at the pediatric surgery department in Cairo University Specialized Pediatric Hospital (Abu EL-Reesh hospital).

Exclusion Criteria:

lung disease cardiac disease Liver disease kidney disease

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
improvement | 6 months
  change of lesion size

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Specialized Pediatric Hospital (Abu EL-Reesh hospital), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No